CLINICAL TRIAL: NCT06896825
Title: Increasing Physical Activity Through Social Support and Stress Resilience (I-PASS) Among Older Adults Living Alone With SCD to Lower ADRD Risk
Brief Title: Increasing Physical Activity Through Social Support and Stress Resilience
Acronym: I-PASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Molly Maxfield, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00020326; 1P30AG086561-01 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Subjective Cognitive Decline (SCD); Sedentary Behavior; Social Isolation in Older Adults
MeSH Terms: conditions — Sedentary Behavior | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tech-enhanced condition (Experimental): Participants in the tech-enhanced condition will receive access to a study specific website (to be developed into an app) and guided use via individual coaching sessions delivered on Zoom. Coaching sessions will align with and reinforce website content, which includes information about the importance of and strategies to increase physical activity, social support, and stress resilience.
  Interventions: Behavioral: Self-monitoring
- Control condition (Active Comparator): Participants in the control condition will receive a study-specific manual containing basic education about the importance of and strategies to increase physical activity, social support, and stress resilience.
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Self-monitoring — All participants will receive a Garmin and use the associated app to monitor their weekly physical activity. Enrolled participants are insufficiently active (engaging in 60 minutes or less of moderate to vigorous physical activity per week) and will receive weekly text messages to incrementally increase physical activity over the course of the study. Goals will be 20% greater than the average daily steps from the previous week, with the ultimate goal of reaching 7000 average daily steps. 7000 average daily steps was selected based on recent findings that it is associated with clinically meaningful health outcomes and being an achievable target for most adults.

SUMMARY:
The goal of this clinical trial is to learn the effects of technology enhancements when combined with basic education, goal-setting, and self-monitoring to increase physical activity among older adults living alone, experiencing subjective cognitive decline, and currently engaging minimal physical activity (60 minutes or less of moderate to vigorous physical activity). Further, we will examine key psychosocial mechanisms believed to contribute to successful promotion of physical activity, which include social support and stress resilience.

The primary questions are to determine whether

* the tech-enhanced condition lead to greater physical activity over time?
* the tech-enhanced condition lead to social support and stress resilience over time?
* social support and stress resilience mediate the relationship between the study condition and physical activity?

All participants will engage in self-monitoring of physical activity, will receive weekly text reminders of their physical activity goals for the week, and will receive basic education about the importance of physical activity, social support, and stress resilience for cognitive, physical, and psychological health. Participants in the tech-enhanced condition will also receive access to a study-specific website and virtual coaching to reinforce the information presented. Researchers will then compare the tech-enhanced condition to the basic education condition to determine the benefits of technology to deliver the intervention materials in order to increase physical activity, social support, and stress resilience.

Participants will:

* Use a Garmin wearable device to monitor their physical activity
* Be randomly assigned to a basic education condition or tech-enhanced condition
* Set achievable goals for weekly physical activity, with incremental increases to achieve 7000 average daily steps by the end of the study
* Respond to surveys to monitor their social support, stress resilience, quality of life, and depression.

The sample has several risk factors for Alzheimer's disease and related dementias: low physical activity, social isolation risk via living alone, and subjective cognitive impairment. Therefore, a long-term goal includes the determination of the intervention's effectiveness at increasing physical activity, social support, and stress resilience to reduce risk for developing dementia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Living alone and community dwelling
* Engaging in 60 minutes or less per week of self-reported moderate-to-vigorous physical activity at screening (based on Exercise Vital Sign Questionnaire)
* Self-reported decline in cognitive functioning
* Self-reported ownership of/willingness to use a smartphone with an iOS or Android operating system (necessary for participants to track their activity using a wearable activity monitor).
* Able to read and speak in English. We hope to offer the intervention in Spanish in the future; however, currently, the study materials are only available in English, and participation will require ability to read and respond to study materials.

Exclusion Criteria:

* Endorsing an item on the Physical Activity Readiness Questionnaire (PAR-Q), unless a physician's note is provided
* Resting blood pressure greater than 200/110 mmHG as assessed at the baseline study assessment (unless a physician's note is provided)
* Plans to relocate out of metropolitan Phoenix, Arizona area in the next 6 months
* Participation in another physical activity, nutrition or weight loss program at time of screening or at any time during the intervention
* Individuals with mild cognitive impairment (MCI), as determined by either a self-report of receiving a diagnosis of MCI from a health care provider or as assessed by the Telephone-Montreal Cognitive Assessment (T-MoCA) at the Baseline Session. A score < 18 is an exclusion criterion.
* Individuals with neurodegenerative (e.g., dementia), developmental (e.g., autism), neurologic (e.g., Parkinson's, epilepsy), or major psychiatric (e.g., bipolar, schizophrenia) diagnoses
* Being previously prescribed one of the 5 approved Alzheimer's medications, including: Donepezil (Aricept), Rivastigmine (Exelon), Galantamine (Razadyne), Memantine (Namenda), Memantine + Donepezil (Namzaric)
* Score of 9 or higher on the 15-item Geriatric Depression Scale (GDS) at the Baseline Session [scores of 9 and higher are indicative of moderate to severe depression]
* Currently taking 2 or more anti-depression medications
* History of stroke
* Incarcerated individuals (i.e., Prisoners)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in accelerometer-measured moderate to vigorous physical activity | One week at baseline and one week after intervention concludes
  ActiGraph GT9X Link Activity monitors worn on non-dominant wrist during waking hours 7 consecutive days will provide objective baseline of moderate to vigorous activity prior to and after the intervention. GTX9X data (collected in raw format) will be aggregated for analysis to epochs of 60 secs or less for comparability to other studies.
Change in Garmin-assessed physical activity | From enrollment to the end of treatment at 3 months
  Participants agree to wear a Garmin throughout the study, offering continuous data about their physical activity. We will use average daily steps (calculated weekly, from Monday to Sunday) to assess physical activity continuously during the intervention.
Change in self-reported physical activity | Reported at baseline and after the 3 month intervention
  Participants will complete an abbreviated 7-Day Physical Activity Recall interview, which assesses self-reported moderate to vigorous physical activity.

SECONDARY OUTCOMES:
Objective Stress Resilience | Assessed at baseline and after the 3 month intervention
  At baseline and 3 months, participants will have blood drawn to assess glial fibrillary acidic protein, an indicator of stress which has also been associated with dementias.
Self-reported stress | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  The 14-item Perceived Stress Scale, with items rated on a 5 point scale (0 to 4). Sum scores are calculated. Possible values range from minimum of 0 to maximum of 56. Higher scores indicate greater perceived stress.
Brief Resilience Scale | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  The 6-item Brief Resilience Scale assesses ability to recover from or adjust to challenges. Items are rated on a 5 point scale. Mean scores are calculated. Possible scores range from a minimum of 1 to a maximum of 5. Higher scores indicating greater resilience.
Social Isolation | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  The 10-item Lubben Social Network Scale assess objective size of social network. Items are rated on a 6 point scale. Sum scores are calculated. Possible scores range from a minimum of 0 and maximum of 60. Higher scores indicate larger social network and contacts.
Self-reported loneliness | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  The 3-item UCLA Loneliness scale assesses the feeling of being alone or lacking companionship. Responses range from 1 to 3. Sum scores are calculated. Possible scores range from a minimum of 3 to a maximum of 9. Higher numbers indicate greater perceived loneliness.
Objective cognitive functioning: Visual memory | Assessed at baseline and after the 3 month intervention
  Participants will complete a visual memory task in which they see a series of pictures in a specified order. Immediately after, they are tasked with placing the pictures in the correct order. This is the Picture Sequence Memory Test from the NIH Toolbox Cognitive Battery. Scoring is automatically calculated by the NIH Toolbox App and is age normed, with higher scores indicating stronger performance on the task.
Objective cognitive functioning: Verbal memory | Assessed at baseline and after the 3 month intervention
  Participants will complete a verbal memory task in which they hear a series of words read and are asked to recall as many as they can immediately after the list; this process is completed three times total to assess both learning and memory. Ten to 15 minutes later, they are asked to recall as many words as possible. This is the Auditory Verbal Learning Test from the NIH Toolbox Cognitive Battery. Scoring is automatically calculated by the NIH Toolbox App and is age normed, with higher scores indicating stronger performance on the task.
Objective cognitive functioning: Executive functioning | Assessed at baseline and after the 3 month intervention
  Participants will complete an executive functioning task requiring set-shifting, or the ability to switch back and forth between multiple aspects of a strategy or task. This is the Dimensional Change Card Sort Task from the NIH Toolbox Cognitive Battery. Scoring is automatically calculated by the NIH Toolbox App and is age normed, with higher scores indicating stronger performance on the task.
Objective cognitive functioning: Processing Speed 1 | Assessed at baseline and after the 3 month intervention
  Participants will complete two tasks assessing processing speed. The first requires visual processing of patterns in two pictures, detecting similarities and differences as quickly as possible without making mistakes. This is the Pattern Comparison Task from the NIH Toolbox Cognitive Battery. Scoring is automatically calculated by the NIH Toolbox App and is age normed, with higher scores indicating stronger performance on the task.
Objective cognitive functioning: Processing Speed 2 | Assessed at baseline and after the 3 month intervention
  Participants will complete two tasks assessing processing speed. The second requires matching of patterns between numbers and symbols as quickly as possible without making mistakes. This is the Oral Symbol Digit Task from the NIH Toolbox Cognitive Battery. Scoring is automatically calculated by the NIH Toolbox App and is age normed, with higher scores indicating stronger performance on the task.
Depression | Assessed at screening and after the 3 month intervention
  Participants will complete the 15-item Geriatric Depression Scale. The items include yes/no responses. Scores will be summed. Possible scores range from a minimum value of 0 to a maximum value of 15. Higher scores indicate greater depression. At eligibility screening, participants must score below 9 on this measure to be included in the study.
General Anxiety | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  Participants will complete the 7-item General Anxiety Disorder Questionnaire. Using a 4 point scale (0 to 3), the items assess worry and anxiety over the past two weeks. Mean scores will be calculated. Possible scores range from a minimum score of 0 to a maximum score of 21. Higher scores indicate greater anxiety.
Health-related quality of life | Assessed at baseline, end of month 1, end of month 2, and end of month 3
  Participants will complete the 4-item health-related quality of life assessment. The items assess self-perceived health and days during the past month they had poor physical health or mental health, and the extent to which poor health kept them from doing daily activities. Mean scores will be calculated. Higher scores indicate poorer health-related quality of life.

OTHER OUTCOMES:
Cognitive Health | Assessed during online eligibility screening and after the 3 month intervention
  To establish eligibility, participants will complete the Telephone administered Montreal Cognitive Assessment (T-MoCA) during the online eligibility screening. Because we are recruiting individuals with subjective cognitive decline, we will rule out potential cognitive impairment with the T-MoCA. Scores are totaled. Possible scores range from 0 to 22. Higher scores indicating better performance. Participants scoring 17 or lower (out of 22) will be ineligible for participation. We will readminister at the end of the 3 month intervention to determine whether change occurred.
Functional Activities | Assessed at baseline and after the 3 month intervention
  Participants will complete the functional activities questionnaire. This measure assesses daily functioning (e.g., preparing meals, managing finances) and participants indicate the level of independence for each. Scores are totaled, with higher scores indicating greater need for support with activities.
Physical Activity Readiness | Assessed at screening and after the 3 month intervention
  During the online eligibility screen, participants will be screened for health-related risks, including risks specific to cardiovascular functioning. This will include administration of the Physical Activity Readiness Questionnaire (PAR-Q+). To ensure participant safety, physician approval and clearance to participate in the intervention will be obtained from participants who report a contraindication to exercise based on the PAR-Q+.
Subjective Cognitive Decline - Eligibility | Assessed at screening and after the 3 month intervention
  During the online eligibility screen, participants will complete the Subjective Cognitive Decline Interview. The experience of subjective cognitive decline is part of the eligibility criteria, so this will be assessed prior to enrollment. In order to be eligible, participants must say yes to the initial question (During the part few years, have you noticed any changes in your mental abilities?) and at least one of the follow up questions (specific to decline in memory, word finding, planning ahead/staying organized, attention, other).
Subjective Cognitive Decline | Assessed at baseline and after the 3 month intervention
  Participants will complete the 20-item Subjective Cognitive Decline questionnaire. They will rate the level of change on a 5 point scale (no change to much worse). Mean scores will be calculated, with higher scores indicating greater perceived decline in cognitive functioning.
Health Status and History | Assessed at baseline and after the 3 month intervention
  Participants will complete a questionnaire assessing previous and current health conditions and status. This questionnaire is adapted from the American College of Sports Medicine's Health History Questionnaire and includes 7 questions. Total scores are not calculated, but individual factors may be examined as covariates (e.g., smoking history, alcohol consumption, etc.)
Demographic information | Assessed at baseline
  Participants will provide basic demographic information. Total scores are not calculated, but individual factors may be examined as covariates (e.g., age, sex, education, etc.)
Family History of Alzheimer's disease and related dementias | Assessed at baseline
  Participants will respond to questions assessing participants' family history of dementia, including parents, siblings, and children. Total scores are not calculated, but family history of dementia may be included as potential covariate for analyses.
Protocol Adherence | Assessed after the 3 month intervention is complete
  To assess protocol adherence, we will calculate number of days the Garmin is worn (all participants), the number of weeks participants met their physical activity goal (all participants), and the number of coaching sessions attended (participants in the tech enhanced group only). Higher numbers for each indicate greater levels of adherence to the protocol.
Treatment Acceptance | Assessed after the 3 month intervention is complete
  To assess overall acceptability of the intervention, participants will complete a treatment acceptance survey specifically adapted for this study. This survey will include satisfaction and acceptability ratings, as well as open-ended questions to obtain participant feedback. Total scores are not calculated. This data will be used to improve the intervention for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Maxfield, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States